CLINICAL TRIAL: NCT01846156
Title: The Best Magnesium Sulphate Protocol for Severe Pre-eclampsia : A Randomized Controlled Trial
Brief Title: New Magnesium Sulphate Protocol for Pre-eclampsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Waleed El-khayat, Assistant Professor of Obstetrics & Gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 52103; 52013 (Registry Identifier: Kasr Aliny)
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Pre-eclampsia
Keywords: convulsion rate
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Abrreviated MgSO4 protocol (Experimental): - Category B : 80 patients given abbreviated doses of MgSO4 (4 grams of MgSO4 on 250 ml ringer solution over 4 hours every 4 hours by IV drip only for 12 hours) in the postpartum period.
  Interventions: Drug: MgSO4
- No maintenance protocol (Experimental): - Category C : 80 patients who will take only loading dose of MgSO4 (6 grams of MgSO4 on 250 ml ringer solutions over 20 minutes) with no postpartum maintenance sulfate
  Interventions: Drug: MgSO4
- standard MgSO4 protocol (Active Comparator): - Category A : 80 patients given full dose of maintenance MgSO4 (4 grams of MgSO4 on 250 ml ringer solution over 4 hours every 4 hours by IV drip for 24 hours) in the postpartum period.
  Interventions: Drug: MgSO4

INTERVENTIONS:
Drug: MgSO4 — A randomized controlled study that compare three regimens for administration of MgSO4 used for the cases of severe pre-eclampsia that will be performed in the Obstetrics & Gynecology Department, Kasr Al-Ainy Hospital, Cairo University

SUMMARY:
there is a standard magnesium sulphate protocol and newer protocols for pre-eclampsia, we need to make a trial to find the best protocol

DETAILED DESCRIPTION:
The aim of our study is to assess the comparative effects of three regimens for the administration of magnesium sulfate when used for the care of women with severe pre-eclampsia.

The study will include 240 pregnant women presenting to the casualty unit with criteria of severe preeclampsia in the form of one of the criteria:-

* Systolic blood pressure ≥ 160.
* Diastolic blood pressure ≥ 110.
* Proteinuria > +2 by dip stick.
* Presence of alarming symptoms (headache, visual disturbance, epigastric pain, vaginal bleeding).
* Fetal growth restriction (IUGR).

After obtaining an informed consent the patients will be subjected to the following:

* Careful history taking including age, parity, gestational age.
* Complete physical examination and assessment of the blood pressure.
* Urine analysis by dipstick.
* All women will take initial MgSO4 (6 grams of MgSO4 on 250 ml ringer solutions over 20 minutes by IV drip) .

Using Random Number Table, the sample size will be divided into three categories:-

* Category A : 80 patients given full dose of maintenance MgSO4 (4 grams of MgSO4 on 250 ml ringer solution over 4 hours every 4 hours by IV drip for 24 hours) in the postpartum period.
* Category B : 80 patients given abbreviated doses of MgSO4 (4 grams of MgSO4 on 250 ml ringer solution over 4 hours every 4 hours by IV drip only for 12 hours) in the postpartum period.
* Category C : 80 patients who will take only loading dose of MgSO4 (6 grams of MgSO4 on 250 ml ringer solutions over 20 minutes) with no postpartum maintenance sulfate.

Inclusion criteria:

* Pregnant females ≥20 weeks of gestation.
* Pregnant females with criteria of severe pre-eclampsia.
* Single or multi-fetal pregnancy.
* Primigravida or Multigravida.

Exclusion criteria:

* Pregnant females < 20 weeks gestation.
* Pregnant females with history of epilepsy.
* Pregnant females with diabetes.
* Pregnant females with chronic hypertension.
* Pregnant females with renal disease.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females ≥20 weeks of gestation.
* Pregnant females with criteria of severe pre-eclampsia.
* Single or multi-fetal pregnancy.
* Primigravida or Multigravida.

Exclusion Criteria:

* Pregnant females < 20 weeks gestation.
* Pregnant females with history of epilepsy.
* Pregnant females with diabetes.
* Pregnant females with chronic hypertension.
* Pregnant females with renal disease.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
duration of MgSo4 treatment | 1 year
  treatment duration

SECONDARY OUTCOMES:
ICU admission | 1 year
  ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-khayat, M.D., Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy hospital, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Derived] Diaz V, Long Q, Oladapo OT. Alternative magnesium sulphate regimens for women with pre-eclampsia and eclampsia. Cochrane Database Syst Rev. 2023 Oct 10;10(10):CD007388. doi: 10.1002/14651858.CD007388.pub3. PMID 37815037